CLINICAL TRIAL: NCT06782789
Title: An Italian Multicentric Retrospective Observational Study to Assess Effectiveness and Safety of the Combination of Tafasitamab and Lenalidomide in Diffuse Large B-cell Lymphoma Patients Treated Under Named Patient Program
Acronym: TALOs
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: TALOs
Record Dates: First submitted 2024-12-03; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-10

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL)
Keywords: tafasitamab; lenalidomide
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study is pilot, observational, retrospective, Italian multicenter study.

DETAILED DESCRIPTION:
The study will involve the collection of patient data from medical records of patients with R/R DLBCL treated with at least one dose of tafasitamab in association with lenalidomide as part of standard of care under the NPP (D.M. 7 Sep 2017), between April 2022 and December 2022, in several selected Italian centres. The observational, non-interventional nature of the study is based on the retrospective observation of current clinical practice without the application of any kind of ad hoc 'intervention' for the study itself. In fact, patients participating in the study will not be subjected to any procedures outside the normal clinical practice; likewise, the clinical variables that will be collected for the study are those that are already commonly collected by the physicians in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of R/R DLBCL.
2. Patientswho received at least one dose of tafasitamab in association with lenalidomide under the NPP (D.M. 7 Sep 2017), between April 2022 and December 2022.
3. Age ≥ 18 years at enrollment.
4. Signature of written informed consent (if applicable).

Exclusion Criteria:

1) R/R DLBCL patients who received tafasitamab in association with lenalidomide in a clinical trial context.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with R/R DLBCL who have received at least one dose of tafasitamab in association with lenalidomide as part of standard of care under the NPP (D.M. 7 Sep 2017), between April 2022 and December 2022.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | through study completion, an average of 2 years
  ORR as the sum of complete response [CR] and partial response [PR] rate. The study aims to retrospectively evaluate the effectiveness of tafasitamab in association with lenalidomide in patients with R/R DLBCL treated with at least one dose of tafasitamab in association with lenalidomide under the NPP.

SECONDARY OUTCOMES:
Duration of Response (DoR) | through study completion, an average of 2 years
  the secondary aim is to evaluate effectiveness of tafasitamab in association with lenalidomide under the NPP (D.M. 7 Sep 2017)
Toxicity of study drug | from enrollment untill 30 days from last infusion
  Type, incidence, severity of any adverse events (AE) occurred from start of treatment to 30 days after last infusion and their possible relationship with study drugs
Progression Free Survival (PFS) | through study completion, an average of 2 years
  The length of time during and after the treatment that patients live with the disease, but it does not get worse. Progression-Free Survival (PFS) will be defined from the date of starting therapy and the date of disease progression, relapse or death from any cause.
Overall Survival (OS) | through study completion, an average of 2 years
  Overall Survival, the percentage of patients alive, is defined from the start date of therapy to the date of death from any cause.
Duration Free Survival (DFS) | through study completion, an average of 2 years
  Disease free survival (DFS) is defined as the time from randomization until evidence of disease recurrence
Best response rate (BRR) | through study completion, an average of 2 years
  Best response rate (BRR)

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (11):
- Italy (11):
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Bologna
  - AO Sant'Anna e San Sebastiano di Caserta, Caserta, Caserta
  - A.R.N.A.S. Garibaldi, Catania, Catania
  - Azienda Ospedaliera Universitaria Arcispedale S. Anna, Ferrara
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Irccs Ospedale San Raffaele, Milan
  - Azienda Ospedaliero-Universitaria Maggiore della Carità, Novara
  - Azienda Ospedaliera Villa Sofia Cervello, Palermo
  - Ospedale Guglielmo da Saliceto di Piacenza, Piacenza
  - IRCCS- Istituto Nazionale Tumori Regina Elena, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma

IPD SHARING:
Plan to Share IPD: No